CLINICAL TRIAL: NCT01176656
Title: Hypoglycemia: Physician and Patient Perspectives
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CUS-DUM-2010/1
Record Dates: First submitted 2010-08-04; First posted 2010-08-06 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Type 2 Diabetes Mellitus; Hypoglycemia
Keywords: Type 2 Diabetes Mellitus; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- SU: T2DM patients with a prescription for a sulfonylurea but no insulin
- Antidiabetic without SU: T2DM patients with an oral antidiabetic drug other than an SU, and no insulin
- Insulin: T2DM patients using insulin, with or without other oral antidiabetics

SUMMARY:
The purpose of this study is to assess the burden of hypoglycemia and identify unmet need related to the management of hypoglycemia among Type 2Diabetes Mellitus (T2DM) patients on OADs and/or insulin. This is an observational study which will identify patients with T2DM in an administrative claims database and will link claims data with results of patient and physician surveys concerning hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* T2DM claims diagnosis (algorithm-based) with at least 2 pharmacy claims for an antidiabetic drug
* at least 1 HbA1c test recorded during the identification period
* continuous enrollment in the health plan for at least 12 months prior to survey date

Exclusion Criteria:

* Type 1 Diabetes Mellitus
* pregnancy or gestational diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with T2DM will be identified from a large U.S. administrative claims database using a claims-based algorithm for T2DM. Patients and their associated physicians will be recruited via mail into the survey portion of this study. Survey results will be linked to actual patient care using the claims records.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
prevalence of hypoglycemia and impact of hypoglycemia | October 2009-October 2010

SECONDARY OUTCOMES:
Patient Reported Outcomes of Hypoglycemia (including fear, awareness, behavioral modification and recovery from hypoglycemia) | October 2009-October 2010
Treatment adherence and modification related to hypoglycemia, including health status, glycemic control and healthcare utilization | October 2009-October 2010

CONTACTS AND LOCATIONS:
Overall Officials: Setareh Williams, PhD, Study Director — AstraZeneca